CLINICAL TRIAL: NCT03422822
Title: A PHASE 3 MULTI-CENTER, LONG-TERM EXTENSION STUDY INVESTIGATING THE EFFICACY AND SAFETY OF ABROCITINIB, WITH OR WITHOUT TOPICAL MEDICATIONS, ADMINISTERED TO SUBJECTS AGED 12 YEARS AND OLDER WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study to Evaluate Efficacy and Safety of PF-04965842 With or Without Topical Medications in Subjects Aged 12 Years and Older With Moderate to Severe Atopic Dermatitis
Acronym: JADE EXTEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451015; JADE EXTEND (Other: Alias Study Number); 2023-508955-37-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT05466578 (Available)
Record Dates: First submitted 2017-12-20; First posted 2018-02-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase; Magnetic Resonance Imaging; MRI
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abrocitinib 100 mg (Experimental): Abrocitinib 100 mg QD PO
  Interventions: Drug: Abrocitinib 100 mg; Drug: Placebo
- Abrocitinib 200 mg (Experimental): Abrocitinib 200 mg QD PO
  Interventions: Drug: Abrocitinib 200 mg; Drug: Abrocitinib 100 mg

INTERVENTIONS:
Drug: Abrocitinib 100 mg — In the initial treatment period, Abrocitinib 100 mg, administered as two tablets to be taken orally once daily.
  Arms: Abrocitinib 100 mg
Drug: Abrocitinib 200 mg — In the initial treatment period, Abrocitinib 200 mg, administered as two tablets to be taken orally once daily.
  Arms: Abrocitinib 200 mg
Drug: Placebo — For subjects whose dose was changed from 100 mg Abrocitinib to placebo, one tablet will be administered to be taken orally once daily for the remainder of the study.
  Arms: Abrocitinib 100 mg
Drug: Abrocitinib 100 mg — For subjects whose dose was changed from 200 mg Abrocitinib to 100 mg PF-04965842, one tablet will be administered to be taken orally once daily for the remainder of the study.
  Arms: Abrocitinib 200 mg
Drug: Abrocitinib 100 mg — In the secondary treatment period, Abrocitinib 100 mg, administered as one tablet to be taken orally once daily.
  Arms: Abrocitinib 100 mg
Drug: Abrocitinib 200 mg — In the secondary treatment period, Abrocitinib 200 mg, administered as two tablets to be taken orally once daily.
  Arms: Abrocitinib 200 mg

SUMMARY:
B7451015 is a Phase 3 study to evaluate Abrocitinib with or without Topical Medications in patients aged 12 years and older who have moderate to severe atopic dermatitis and have completed a qualifying parent study. The efficacy and safety of two dosage strengths of Abrocitinib, 100 mg and 200 mg taken orally once daily, will be evaluated over variable lengths of study participation. The study consists of a 92 week initial treatment period followed by a variable length secondary treatment period during which subjects will receive treatment with open-label abrocitinib until availability of commercial product in their country, or until the sponsor terminates the study in that country.

The B7451015 study also includes a sub-study evaluating whether abrocitinib has any potential effects on adolescent bone with regard to abnormal bone findings in knee MRI. The sub-study will be conducted in selected countries at selected sites. Eligible subjects are those who were 12 to <18 years of age at the screening visit of the qualifying parent study and who are currently participating in the main B7451015 study. The sub-study will include serial Magnetic Resonance Imaging (MRI) annually and continue until all enrolled subjects are 18 years of age and have been imaged at least once or have discontinued/withdrawn.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject or their parent(s)/legal guardian, if applicable, have been informed of all pertinent aspects of the study.
2. Male or female subjects of 12 years of age or older, at the time of informed consent and meets inclusion criterion for minimum body weight (if applicable) from qualifying Parent study. Adolescent subjects below the age of 18 years old (or country-specific age of majority) will only be enrolled in this study if instructed by the sponsor and approved by the country or regulatory/health authority. If these approvals have not been granted, only subjects aged 18 years (or country-specific age of majority) and older will be enrolled.
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
4. Must have completed the full treatment period of a qualifying Parent study OR must have completed the full rescue treatment period of a qualifying Parent study (if applicable) OR must have completed the full open-label run-in period in B7451014 and did not meet the protocol-specified response criteria at Week 12.
5. Female subjects who are of childbearing potential (which includes all female subjects aged 12 years and older, regardless of whether they have experienced menarche) must ot be intending to become pregnant, currently pregnant, or lactating. The following onditions apply:

   1. Female subjects of childbearing potential must have a confirmed negative pregnancy test prior to allocation to treatment.
   2. Female subjects of childbearing potential must agree to use a highly effective method of contraception (as per Section 4.4.1) for the duration of the active treatment period and for at least 28 days after the last dose of investigational product.

For Czech Republic only, 5 b. is revised and 5 c. is added to require:

Female subjects of childbearing potential 15 years of age who are at risk of pregnancy must agree to use a highly effective method of contraception for the duration of the active treatment period and for at least 28 days after the last dose of investigational product.

c. Female subjects less than 15 years of age must not be sexually active, and abstinence per the below definition should be confirmed prior to enrollment. NOTE: Sexual abstinence, defined as completely and persistently refraining from all heterosexual intercourse (including during the entire period of risk associated with the study treatments) may obviate the need for contraception ONLY if this is the preferred and usual lifestyle of the subject.

6. Female subjects of non-childbearing potential must meet at least 1 of the following criteria:

1. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
2. Have medically confirmed ovarian failure; or
3. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential. 7. Must agree to avoid prolonged exposure to the sun and not to use tanning booths, sun lamps or other ultraviolet light sources during the study.

   8. Must agree to avoid use of prohibited medications throughout the duration of the study. Exclusion Criteria
   1. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
   2. Currently have active forms of other inflammatory skin diseases, ie, not AD or have evidence of skin conditions (eg, psoriasis, seborrheic dermatitis, Lupus) at the time of Day -1 that would interfere with evaluation of atopic dermatitis or response to treatment.
   3. Discontinued from treatment (or rescue treatment period/open-label run-in period, if applicable) early in a qualifying Parent study OR triggered a discontinuation criterion at any point during the qualifying Parent study which in the opinion of the investigator, or sponsor, is an ongoing safety concern.
   4. Ongoing adverse event in the qualifying Parent study which in the opinion of the investigator, or sponsor, is an ongoing safety concern.
   5. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.

   There are also additional separate inclusion and exclusion criteria to assess eligibility specifically for the B7451015 MRI sub-study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3166 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  The incidence of treatment emergent adverse events
Serious adverse events and adverse events leading to discontinuation | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  The incidence of serious adverse events and adverse events leading to discontinuation
Change from baseline in clinical laboratory values | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Change from baseline in clinical laboratory values
Change from baseline in electrocardiogram (ECG) measurements | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Change from baseline in electrocardiogram (ECG) measurements
Change from baseline in vital signs | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Change from baseline in vital signs

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | Baseline, Week 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
  Response based on the IGA score of clear (0) or almost clear (1) (on a 5 point scale) and a reduction from baseline of >=2 points at all scheduled time points
Eczema Area and Severity Index (EASI) | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Response based on greater than or equal to 50%, 75% and 90% improvement from baseline in the EASI total score (EASI50, EASI75, and EASI90) at all scheduled time points
Pruritus Numerical Rating Scale (NRS) | Baseline, Week 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
  Response based on an improvement greater than or equal to 3 points and greater than or equal to 4 points from baseline in the pruritus NRS at all scheduled time points
Patient Global Assessment (PtGA) | Baseline, Week 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
  Change from baseline of PtGA at all scheduled time points
Body Surface Area (BSA) affected | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Change from baseline in the percentage BSA affected at all scheduled time points
Dermatology Life Quality Index (DLQI) or Children's DLQI (CDLQI) | Baseline, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
  Change from baseline in DLQI or CDLQI at all scheduled time points
Patient Oriented Eczema Measure (POEM) | Baseline, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 92
  Change from baseline in POEM at all scheduled time points
Hospital Anxiety and Depression Scale (HADS) | Baseline, Week 12, Week 24, Week 36, Week 48, Week 60, Week 64, Week 72, Week 84, Week 92, Week 96
  Change from baseline in HADS at all scheduled time points
EuroQol Quality of Life 5 Dimension 5 Level Scale (EQ-5D-5L) or EuroQol Quality of Life 5 Dimension Youth Scale (EQ-5D-Y) | Baseline, Week 24, Week 48, Week 60, Week 72, Week 92
  Change from baseline of EQ-5D-5L or EQ-5D-Y at all scheduled time points
Steroid-Free Days | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Number of steroid-free days will be assessed throughout the duration of the study.
Serum Hs-CRP Levels | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Serum Hs-CRP levels at all scheduled time points
Change in height standard deviation score (SDS) | Throughout study regardless of availability of commercial product until at least 2024, or until the sponsor terminates the study; an estimated maximum of 8 years
  Change in height standard deviation score (SDS) at all scheduled time points
Proportion of abnormal findings in knee MRI in adolescent subjects exposed to abrocitinib 100mg and 200mg QD | Throughout sub-study until all enrolled subjects are 18 years of age and have been imaged at least once or have discontinued or withdrawn; an estimated maximum of 4 years
  Proportion of abnormal findings in knee MRI in adolescent subjects exposed to abrocitinib 100mg and 200mg QD

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (536):
- United States (154):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham - Dermatology Research Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham Hospital Outreach Lab, Birmingham, Alabama
  - The University of Alabama at Birmingham, Department of Dermatology, Birmingham, Alabama
  - Emmaus Research Center, Inc., Anaheim, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Marvel Research, LLC, Huntington Beach, California
  - Tilda Research Inc., Irvine, California
  - Beach Allergy and Asthma Specialty Group, A Medical Corporation, Long Beach, California
  - Keck School of Medicine of University of Southern California, Los Angeles, California
  - Wallace Medical Group, Inc, Los Angeles, California
  - Allergy & Asthma Associates of Southern California dba Southern California Research, Mission Viejo, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Peninsula Headlands LLC, Rolling Hills Estates, California
  - UC Davis Health, Sacramento, California
  - MedDerm Associates, San Diego, California
  - University of California San Diego Dermatology, San Diego, California
  - Synergy Dermatology, San Francisco, California
  - San Luis Dermatology and Laser Clinic, San Luis Obispo, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Wolverine Clinical Trials, Llc, Santa Ana, California
  - Mosaic Dermatology, Santa Monica, California
  - Clinical Science Institute, Santa Monica, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Colorado Springs Dermatology Clinic, PC, Colorado Springs, Colorado
  - Skin Care Research, Boca Raton, Florida
  - Renaissance Research and Medical Group, Inc, Cape Coral, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Homestead Research Institute, Homestead, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - C & R Research Services USA, Inc, Kendall, Florida
  - Clinical Trials Solutions, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - Suncoast Research Associates, Miami, Florida
  - La Salud Research Clinic, Inc., Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - South Miami Medical & Research Group, Inc., Miami, Florida
  - Ciocca Dermatology, PA, Miami, Florida
  - Miami Dermatology & Laser Research, LLC, Miami, Florida
  - INTERMED Medical Research Center, Inc, Miami, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Wellness Clinical Research, LLC, Miami Lakes, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Pediatric Dermatology Orlando, Orlando, Florida
  - Advent Health Orlando - Investigational Drug Services, Orlando, Florida
  - Outpatient Services Center - AdventHealth Orlando, Orlando, Florida
  - Pediatric Outpatient Procedures and Sedation, Orlando, Florida
  - Accel Research Sites - Nona Pediatric Center, Orlando, Florida
  - Olympian Clinical Research, St. Petersburg, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - University of South Florida; Asthma, Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Integrated Clinical Research, West Palm Beach, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - IACT Health, Columbus, Georgia
  - One Health Research Clinic Atlanta, LLC, Johns Creek, Georgia
  - Dermatologic Surgery Specialists, PC, Macon, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - ASR, LLC, Nampa, Idaho
  - Midwest Allergy Sinus Asthma, SC, Normal, Illinois
  - NorthShore University HealthSystem - Dermatology, Skokie, Illinois
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Ds Research, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Qualmedica Research, LLC., Owensboro, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - DermAssociates, LLC, Rockville, Maryland
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Clinical Unit for Research Trials in Skin (CURTIS), Boston, Massachusetts
  - MetroBoston Clinical Partners, LLC, Brighton, Massachusetts
  - Clarkston Skin Research, Clarkston, Michigan
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - Onyx Clinical Research, Flint, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Henry Ford Medical Center - Farmington Road, West Bloomfield, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Saint Louis University Dermatology, St Louis, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UR Dermatology Clinical Trials Unit at College Town, Rochester, New York
  - Investigational Drug Service, Rochester, New York
  - Cary Dermatology Center, PA, Cary, North Carolina
  - Accellacare - Cary, Cary, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - M3-Wake Research, Inc., Raleigh, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Winston-Salem Dermatology and Surgery Center, PLLC, Winston-Salem, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio State University Dermatology East, Gahanna, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Portland Clinical Research dba Columbia Asthma & Allergy Clinic, Clackamas, Oregon
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - MUSC SCTR Research Nexus Clinic and Laboratory, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Tanenbaum Dermatology Center, Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - The University of Texas Health Science Center Houston, Bellaire, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Ventavia Research Group, Hurst, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Center for Clinical Studies, LTD.LLP, Webster, Texas
  - Summit Clinical Research, LLC, Franklin, Virginia
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
  - Fort Norfolk Diagnostic Center, Norfolk, Virginia
  - Pace Dermatology Associates, Lakewood, Washington
  - Dermatology Associates of Seattle, Seattle, Washington
  - Dermatology Specialists of Spokane, Spokane, Washington
  - Principle Research Solutions, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - Multicare Institute for Research and Innovation, Tacoma, Washington
  - Pace Dermatology Associates, Tacoma, Washington
  - Children's Hospital of Wisconsin Investigational Drug Service, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin Translational Research Unit, Milwaukee, Wisconsin
- Argentina (6):
  - CONEXA Investigación Clínica S.A., CABA, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Servicio de Investigacion de Patolog-ias Alergicas del Instituto ABC - Rosario, Rosario, Santa Fe Province
  - Psoriahue Medicina Interdisciplinaria, C.a.b.a.
  - CINME Centro de Investigaciones Metabolicas, C.a.b.a
- Australia (16):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - St George Dermatology & Skin Cancer Centre, Kogarah, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Skin Hospital, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - North Eastern Health Specialists, Campbelltown, South Australia
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Skin Health Institute Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Emeritus Research, Camberwell
  - Royal Melbourne Hospital, Parkville
  - Royal North Shore Hospital, Saint Leonards NSW
- Belgium (3):
  - University Hospital Brussels, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Antwerp, Edegem
- Brazil (8):
  - Instituto de Dermatologia e Estética do Brasil LTDA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul
  - Associacao dos Funcionarios Públicos do Estado do Rio Grande do Sul - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Fundacao do ABC - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Tecnolab Medicina Diagnostica, Santo André, São Paulo
  - Pesquisare Saude S/S Ltda, Santo André, São Paulo
  - Tecnolab - Unidade Matriz, São Bernardo do Campo, São Paulo
  - IBPClin Pesquisa Clinica, Rio de Janeiro
- Bulgaria (13):
  - MHAT Dobrich AD, Dobrich
  - MC Asklepii" OOD, Dupnitsa
  - MHAT ''Dr. Tota Venkova'' AD, Gabrovo
  - "Acibadem City Clinic MHAT Tokuda" EAD, Sofia
  - "DCC Aleksandrovska" EOOD, Sofia
  - "DCC Fokus-5-Medical Establishment for OutpatientCare"EOOD, Sofia
  - Military Medical Academy MHAT Sofia, Sofia
  - Dermatology Clinic "Sofia" - group practice for specialized outpatient medical care, Sofia
  - "Mc Synexus Sofia" Eood, Sofia
  - ACIBADEM City Clinic Diagnostic-Consultative Center EOOD, Sofia
  - Medical Center Synexus Sofia EOOD-branch Stara Zagora, Stara Zagora
  - "ACIBADEM City Clinic Medical Center Varna" EOOD, Varna
  - "DCC Mladost-M Varna" OOD, Varna
- Canada (40):
  - Dermatology Research Institute, Calgary, Alberta
  - Beacon Dermatology, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - CARE Clinic Ltd, Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc, Surrey, British Columbia
  - University of British Columbia Department of Dermatology and Skin Science, Vancouver, British Columbia
  - Pacific Dermaesthetics Inc., Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Karma Clinical Trials, Inc., St. John's, Newfoundland and Labrador
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - Derm Effects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - Oshawa Clinic Dermatology Trials, Oshawa, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - North York Research Inc., Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Research Toronto, Toronto, Ontario
  - AvantDerm, Toronto, Ontario
  - Manna Research Inc.(Toronto), Toronto, Ontario
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Clinique de Radiologie du Saguenay Enr., Chicoutimi, Quebec
  - Intermed groupe santé, Chicoutimi, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Dr. Rachel Asiniwasis, Medical Professional Corp., Regina, Saskatchewan
  - Centre de Recherche Saint-Louis inc., Québec
- Chile (6):
  - Centro Medico SkinMed Limitada, Santiago, Santiago Metropolitan
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
  - CEC Spa, Santiago, Santiago Metropolitan
  - MIRES (M Y F Estudios Clínicos Limitada), Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
- China (25):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The second Xiangya Hospital,Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Dermatological department, Changsha, Hunan
  - The First Affiliated Hospital With Nanjing University, Nanjing, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Provincial Institute of Dermatology and Venereology & Shandong Provincial Hospital for Skin, Jinan, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Dermatological Department, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University School of Medicine/Dermatology and STD Dept, Hangzhou, Zhejiang
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine/Dermatology Dept, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital/Dermatology Department, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Army Medical University,PLA, Chongqing
  - Dermatology Department, Shanghai Changzheng Hospital, Shanghai
  - Xin Hua Hospital Affiliated to Shanghai Jiaotong University School of Medicine/Dermatology, Shanghai
  - Shanghai Dermatology Hospital, Shanghai
- Czechia (21):
  - Lekarna Pod Kankem, Kunta Hora
  - Kozni ambulance Kutna Hora, s.r.o, Kutná Hora
  - Dermamedica S.R.O., Náchod
  - Lekarna U Stribrneho orla (Pharmacy), Náchod
  - CCR Ostrava, s.r.o., Ostrava
  - Lekarna Rezidence Nova Karolina, Ostrava
  - Apavar Lekarna, Ostrava
  - Lekarna Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni Nemocnice Ostrava, Kozni oddeleni, Ostrava - Poruba
  - BENU Lekarna, Pardubice
  - PRATIA Pardubice a.s., Pardubice
  - Lekarna, Nemocnice Pardubickeho kraje, a.s. , Pardubicka nemocnice, Pardubice
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
  - Lekarna Pod Platany (Pharmacy), Prague
  - Prof. MUDr.Petr Arenberger, DrSc. MBA, Prague
  - Lekarna U Spasitele, Prague
  - PRATIA Prague s.r.o., Prague
  - Dermatovenerologicka ambulance, Svitavy
  - Lekarna na Hranicni (Pharmacy), Svitavy
  - Krajska zdravotni a.s., Masarykova nemocnice o.z., Ústí nad Labem
  - Lekarna Masarykovy nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Finland (3):
  - Terveystalo Tampere, Tampere
  - Mehiläinen Neo, Turku
  - Turun yliopistollinen keskussairaala, Turku
- Germany (28):
  - Dermazentrum Augsburg, Augsburg
  - Licca Clinical Research Institute, Augsburg
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Hautzentrum Friedrichshain Studien, Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA GmbH, Berlin
  - Klinikum Bielefeld Rosenhoehe, Bielefeld
  - Universitaetsklinikum Bonn, Bonn
  - Klinische Forschung Dresden GmbH, Dresden
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - IKF Pneumologie GmbH & Co KG; Institut für klinische Forschung, Frankfurt
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Klinische Forschung Hamburg GmbH, Hamburg
  - MENSINGDERMA research GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Praxis Dr. med. Beate Schwarz, Langenau
  - Velocity Clinical Research Germany GmbH, Leipzig
  - Universitaetsklinikum Schleswig-Holstein, Campus Luebeck, Lübeck
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - Universitätsklinikum Marburg, Marburg
  - Ludwig-Maximilians-University Munich, Munich
  - University of Muenster, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Hautaerztliche Gemeinschaftspraxis Dres. Leitz und Kollegen, Stuttgart
- Hungary (15):
  - Clinexpert Kft., Budapest
  - SE AOK Bor, Nemikortani es Boronkologiai Klinika, Budapest
  - Bp. Főváros XIX. Kerület Önkormányzat Kispesti Eü. Intézete, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Kft., Encs
  - Bugát Pál Kórház, Bőrgyógyászati Szakrendelés, Gyöngyös
  - Trial Pharma Kft., Győr
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. Synexus Gyula DRS, Gyula
  - Trial Pharma Kft., Kaposvár
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Gyermek Gasztroenterológia II. emelet, Miskolc
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Bor-,Nemikortani es Onkodermatologiai Klinika, Pécs
  - Trial Pharma Kft., Püspökladány
  - Szegedi Tudomanyegyetem Szent-Györgyi Albert, Szeged
  - ALLERGO-DERM BAKOS Kft., Szolnok
  - Medmare Bt, Veszprém
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - AOU Policlinico Sant'Orsola Malpighi, Bologna, BO
  - Universita degli Studi G. D'Annunzio -CeSi-MeT, Chieti, CH
  - Ospedale Policlinico San Martino, Genova, GE
  - AOU Policlinico di Modena Struttura complessa di Dermatologia, Modena, MO
  - Istituto Clinico Humanitas IRCSS - UOC di Dermatologia, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - IFO lstituto Dermatologico San Gallicano IRCCS, Roma
  - Universita del Sacro Cuore, Policlinico Agostino Gemelli, Istituto Di Dermatologia, Rome
- Japan (16):
  - Kawashima Dermatology Clinic, Ichikawa, Chiba
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Dermatology Shimizu Clinic, Kobe, Hyōgo
  - Queen's square Medical Facilities Queen's square Dermatology and Allergology, Yokohama, Kanagawa
  - Noguchi Dermatology Clinic, Kamimashiki-gun, Kumamoto
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Iidabashi Skin Clinic, Chiyoda-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Matsuyama Dermatology Clinic, Nakano-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjyuku-ku, Tokyo
  - Hoshikuma Dermatology・Allergy Clinic, Fukuoka
  - Matsuda Tomoko Dermatological Clinic, Fukuoka
  - Sanrui Hifuka, Saitama
- Latvia (7):
  - Riga 1st Hospital, Clinic of Dermatology and STD, Riga
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Health Centre 4 Ltd. Diagnostics Centre, Riga
  - Childrens Clinical University Hospital State SLLC, Riga
  - Health and Aesthetics Ltd, Riga
  - Health Centre 4 Ltd, Dermatology Clinics, Riga
  - Outpatient Clinic Of Ventspils, Ventspils
- Mexico (17):
  - Clinical Research Institute S.C., Saltillo, Coahuila
  - Hospital Infantil de Mexico Federico Gomez, Del. Cuauhtemoc, Mexico City
  - JM Research SC, Cuernavaca, Morelos
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Unidad de Atención Médica e Investigación en Salud, Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Derma Norte del Bajio S.C., Aguascalientes
  - Centro de Investigacion Integral MEDIVEST, S.C., Chihuahua City
  - Servicios Hospitalarios de Mexico S.A. de C.V. (Hospital Ángeles Chihuahua), Chihuahua City
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
  - Hospital de Jesus, I.A.P., Mexico City
  - Cryptex Investigación Clínica, S.A. de C.V., Mexico City
  - Arke Estudios Clinicos Sa De Cv, Mexico City
  - Trials in Medicine S.C., Mexico City
  - Eukarya Pharmasite S.C., Monterrey
  - SMIQ, S. de R. L. de C.V., Querétaro
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- Universitair Medisch Centrum (UMC) Utrecht, Utrecht, Netherlands
- Poland (57):
  - NZOZ Specjalistyczny Osrodek Dermatologiczny DERMAL s.c., Bialystok
  - KLIMED Marek Klimkiewicz, Bialystok
  - Clinica Dermatoestetica Prywatny Gabinet Dermatologiczny i Alergologiczny, Bydgoszcz
  - DERMAPOLIS Medical Dermatology Center dr n. med. Edyta Gębska, Chorzów
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - Uniwersyteckie Centrum Kliniczne Klinika Dermatologii, Wenerologii i Alergologii, Gdansk
  - Neutrum Lekarze M. Hlebowicz i Partnerzy Spolka Partnerska, Gdansk
  - Szpital Sw. Wojciecha, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - MCBK, Grodzisk Mazowiecki
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - MULTIKLINIKA Salute Sp. z o.o., Katowice
  - Silmedic Sp. z o.o., Oddzial w Katowicach, Katowice
  - Care Clinic Centrum Medyczne, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Pro Familia Altera Sp. z o.o., Katowice
  - Gabinet Dermatologiczny Beata Krecisz, Kielce
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Badan Klinicznych JCI, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Centrum Nowoczesnych Terapii "DOBRY LEKARZ" sp. z o.o., Krakow
  - AWP Klinika Dermatologii Pod Fortem Anna Wojas-Pelc, Krakow
  - Centrum Medyczne Promed, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Prywatna Praktyka Lekarska - Adam Smialowski INTERMED KSAWEROW, Ksawerów
  - NZOZ "DERMED" Centrum Medyczne Sp. z o.o. - Oddzial w Lodzi, Lodz
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Osrodek badan klinicznych AppleTree Clinics, Lodz
  - Dermoklinika-Centrum Medyczne s.c. M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - NZOZ "Med-Laser" Borzecki Spolka Jawna, Lublin
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan
  - Clinical Research Center Sp. z o.o. MEDIC-R Sp. k., Poznan
  - Gabinety Lekarskie Rivermed, Poznan
  - LIFT-MED Spolka Akcyjna, Rybnik
  - Kliniczny Szpital Wojewodzki nr 1 im. F. Chopina, Klinika Dermatologii, Rzeszów
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów
  - Andrzej Krolicki, Tomasz Kochanowski "Laser Clinic" S.C., Szczecin
  - Twoja Przychodnia Szczecinskie Centrum Medyczne, Szczecin
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z o.o., Tarnów
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji w Warszawie, Warsaw
  - RCMed Oddzial Warszawa, Warsaw
  - Carpe Diem Centrum Medycyny Estetycznej, Warsaw
  - REUMATIKA - "Centrum Reumatologii" NZOZ 2, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - ETG Warszawa, Warsaw
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - Wojskowy Instytut Medyczny, Klinika Dermatologiczna, Warsaw
  - EMC Instytut Medyczny S.A. Przychodnia przy ul. Lowieckiej, Wroclaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Lukasz Matusiak "4Health", Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Kliniczny Oddzial Chorob Wewnetrznych, Dermatologii i Alergologii, Zabrze
- Romania (3):
  - SC Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov, JUD. Brasov
  - Cabinet Medical de Dermatovenerologie Prof. Dr. Orasan Remus Ioan, Cluj-Napoca, JUD. CLUJ
  - SC Delta Health Care SRL, Bucharest
- Russia (14):
  - SBIH "Chelyabinsk Regional Clinical Dermatovenerology dispensary", Chelyabinsk
  - Limited Liability Company "Medical Center "Rheuma-Med", Kemerovo
  - Clinic of FSBEI HE Kirov SMU MOH Russia, Kirov
  - FSBI "State Research Centre of Dermatovenereology and Cosmetology" MoH RF, Moscow
  - NRC Institute of Immunology FMBA of Russia, Moscow
  - SBI RR "Skin and Venereal Dispensary", Rostov-on-Don
  - SBI RR "Regional Clinical Skin and Veneral Dispensary", Ryazan
  - LLC "Pierre Wolkenstein Clinic of Skin Diseases", Saint Petersburg
  - Vitiligo center, Saint Petersburg
  - FSBEI HE "St. Petersburg State Pediatric Medical University" MoH RF, Saint Petersburg
  - Limited Liability Company "Sanavita", Saint Petersburg
  - "Medical Research Institute", LLC, Saint Petersburg
  - FSBEI HE I.P.Pavlov SPbSMU MOH Russia, Saint Petersburg
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
- Serbia (3):
  - Military Medical Academy, Belgrade
  - Clinical Centre Nis, Niš
  - General Hospital Pancevo, Pančevo
- Slovakia (9):
  - Narodny ustav detskych chorob, Bratislava
  - BeneDerma s.r.o., Bratislava
  - Derma therapy spol. s.r.o, Dermatovenerologicka ambulancia, Bratislava
  - Summit Clinical Research, s.r.o., Bratislava - Mestská Cast Nove Mesto
  - SKINKLINIK s.r.o., Bratislava- Mestská Časť Nové Mesto
  - Nemocnica Kosice-Saca, a.s., 1. sukromna nemocnica, Kozna ambulancia, Kosice-Saca
  - Derma-beauty, s.r.o., Dermatovenerologicka ambulancia, Nitra
  - Fakultna nemocnica s poliklinikou Nove Zamky, Dermatovenerologicka klinika, Nové Zámky
  - SANARE spol.s.r.o., Svidník
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital CNUH, Daejeon
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei Univ. Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (20):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau Servicio de Dermatologia, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital del Nino Jesus, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro de Especialidades Mollabao (Area Sanitaria de Pontevedra e O Salnes), Pontevedra
  - Hospital de Montecelo, Pontevedra
  - Hospital Universitario Virgen de la Macarena, Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (9):
  - Taipei Veterans General Hospital, Taipei, Taiwan (r.o.c)
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan
- United Kingdom (18):
  - Medinova Research, Wokingham, Berkshire
  - MeDiNova West London Quality Research Sites, Wokingham, Berkshire
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth, Devon
  - Royal free London NHS Foundation Trust, London, Greater London
  - MeDiNova South London Quality Research Site, Orpington, KENT
  - Accellacare North London, Northwood, Middlesex
  - Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire
  - Sheffield Children's NHS Foundation Trust, Sheffield, South Yorkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Northern General Hospital, Sheffield, South Yorkshire
  - MAC Clinical Research, Blackpool
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - MAC Clinical Research, Cannock
  - Accellacare Warwickshire, Coventry
  - West Glasgow Ambulatory Care Hospital, Glasgow
  - Guy's Hospital-Guy's and St Thomas NHS Foundation Trust, London
  - MAC Clinical Research Ltd, Manchester
  - Accellacare South London, Orpington
  - Accellacare Yorkshire, Shipley

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paller AS, Eichenfield LF, Irvine AD, Flohr C, Wollenberg A, Barbarot S, Bangert C, Spergel JM, Selfridge A, Biswas P, Fan H, Alderfer J, Watkins M, Koppensteiner H. Integrated Efficacy and Safety Analysis of Abrocitinib in Adolescents With Moderate-to-Severe Atopic Dermatitis. Allergy. 2025 Aug;80(8):2213-2224. doi: 10.1111/all.16512. Epub 2025 Mar 3. PMID 40028832
- [Derived] Silverberg JI, Simpson EL, Pink AE, Weidinger S, Chan G, Biswas P, Clibborn C, Guler E. Switching from Dupilumab to Abrocitinib in Patients With Moderate-to-Severe Atopic Dermatitis: A Post Hoc Analysis of Efficacy After Treatment With Dupilumab in JADE DARE. Dermatol Ther (Heidelb). 2025 Feb;15(2):367-380. doi: 10.1007/s13555-024-01320-y. Epub 2025 Feb 4. PMID 39903335
- [Derived] Silverberg JI, Thyssen JP, Lazariciu I, Myers DE, Guler E, Chovatiya R. Abrocitinib may improve itch and quality of life in patients with itch-dominant atopic dermatitis. Skin Health Dis. 2024 May 5;4(4):e382. doi: 10.1002/ski2.382. eCollection 2024 Aug. PMID 39104653
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451015